CLINICAL TRIAL: NCT06453044
Title: A Phase 2 Study of Mosunetuzumab With Polatuzumab Vedotin in Patients With Relapsed/Refractory Follicular Lymphoma
Brief Title: Mosunetuzumab and Polatuzumab Vedotin for the Treatment of Patients With Relapsed or Refractory Grade 1-3a Follicular Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23003; NCI-2024-04429 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23003 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2024-05-30; First posted 2024-06-11 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3a Follicular Lymphoma; Refractory Grade 1 Follicular Lymphoma; Refractory Grade 2 Follicular Lymphoma; Refractory Grade 3a Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Specimen Handling; Magnetic Resonance Spectroscopy; polatuzumab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (mosunetuzumab, polatuzumab vedotin) (Experimental): Patients receive polatuzumab vedotin IV over 30-90 minutes on day 1 of each cycle. Cycles repeat every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive mosunetuzumab SC on days 1, 8 and 15 of cycle 1 and day 1 of remaining cycles. Cycles repeat every 21 days for up to 8-17 cycles in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection and CT, PET/CT, or MRI throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Biological: Mosunetuzumab; Drug: Polatuzumab Vedotin; Procedure: Positron Emission Tomography; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Mosunetuzumab — Given SC
  Other Names: Anti-CD20 x Anti-CD3 Bispecific Monoclonal Antibody BTCT4465A; BTCT 4465A; BTCT-4465A; BTCT4465A; CD20/CD3 BiMAb BTCT4465A; Lunsumio; Mosunetuzumab-axgb; RG 7828; RG-7828; RG7828; RO7030816
Drug: Polatuzumab Vedotin — Given IV
  Other Names: ADC DCDS4501A; Antibody-Drug Conjugate DCDS4501A; DCDS4501A; FCU 2711; polatuzumab vedotin-piiq; Polivy; RG7596; Ro 5541077-000
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Other: Questionnaire Administration — Ancillary Studies

SUMMARY:
This phase II trial tests how well mosunetuzumab and polatuzumab vedotin works in treating patients with grade 1-3a follicular lymphoma that has come back after a period of improvement (relapsed) or that has not responded to previous treatment (refractory). Mosunetuzumab is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. Polatuzumab vedotin is a monoclonal antibody, polatuzumab, linked to a toxic agent called vedotin. Polatuzumab attaches to CD79B positive cancer cells in a targeted way and delivers vedotin to kill them. Giving mosunetuzumab and polatuzumab vedotin may kill more cancer cells in patients with relapsed or refractory grade 1-3a follicular lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the safety and tolerability of mosunetuzumab plus polatuzumab vedotin in patients with relapsed/refractory (R/R) follicular lymphoma (FL). (Safety lead-in) II. Estimate the complete response (CR) rate to mosunetuzumab plus polatuzumab vedotin in R/R FL patients. (Phase II)

SECONDARY OBJECTIVES:

I. Estimate the overall response rate (ORR), time to first CR, time to best response, duration of response (DOR), duration of response among CR (DORC), progression-free survival (PFS), overall survival (OS), and quality of life (QOL) in R/R FL patients treated with mosunetuzumab plus polatuzumab vedotin.

II. Evaluate the toxicity of mosunetuzumab plus polatuzumab vedotin for R/R FL. III. Examine the use of tocilizumab for cytokine release syndrome (CRS) in R/R FL patients treated with mosunetuzumab plus polatuzumab vedotin.

EXPLORATORY OBJECTIVES:

I. Assess baseline and on-treatment biomarkers, and evaluate association with anti-tumor activity and safety.

II. Examine the type and incidence of CD20 gene mutations/ downregulation at relapse in R/R FL patients treated with mosunetuzumab plus polatuzumab vedotin.

OUTLINE:

Patients receive polatuzumab vedotin intravenously (IV) over 30-90 minutes on day 1 of each cycle. Cycles repeat every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive mosunetuzumab subcutaneously (SC) on days 1, 8 and 15 of cycle 1 and day 1 of remaining cycles. Cycles repeat every 21 days for up to 8-17 cycles in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection and computed tomography (CT), positron emission tomography (PET)/CT, or magnetic resonance imaging (MRI) throughout the study.

After completion of study treatment, patients are followed up at 30 days and then for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Be willing to provide tissue from a fresh core or excisional biopsy (performed as standard of care) of a tumor lesion prior to starting study therapy or from diagnostic tumor biopsies

  * If unavailable, exceptions may be granted with study principal investigator (PI) approval
* Age: ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) ≤ 2
* Histologically confirmed diagnosis of follicular lymphoma grade 1-3a according to the World Health Organization (WHO) classification. Note: A history of diffuse large B-cell lymphoma (DLBCL) and/or grade 3b follicular lymphoma is allowed (follicular large B-cell lymphoma in the WHO 5th classification of mature B-cell lymphoma) but these cannot be present at the time of study enrollment. Enrollment of any such cases on this study must receive prior approval by the study PI
* Relapsed/ refractory disease after at least one prior line of therapy. Relapse must have been confirmed histologically
* Tumor must be positive for CD20 by immunohistochemistry or flow cytometry after the most recent therapy. Note: As a pan-B marker, CD79B+ is nearly always present and is not a criterion for inclusion
* Active disease requiring treatment per treating physician's decision
* Radiographically measurable disease by Lugano criteria (e.g., one or more nodal sites of disease ≥ 1.5 cm and/or at least one extranodal site of disease ≥ 1.0 cm in longest dimension)
* Fully recovered from the acute toxic effects (except alopecia) to ≤ grade 1 to prior anti-cancer therapy
* WITHOUT BONE MARROW INVOLVEMENT BY LYMPHOMA: Absolute neutrophil count (ANC) ≥ 1,000/mm^3. NOTE: Growth factor is not permitted within 7 days of ANC assessment unless cytopenia is secondary to disease involvement
* WITH BONE MARROW INVOLVEMENT BY LYMPHOMA AND/OR DISEASE-RELATED NEUTROPENIAS: ANC ≥ 500/mm^3. NOTE: Growth factor is not permitted within 7 days of ANC assessment unless cytopenia is secondary to disease involvement
* WITHOUT BONE MARROW INVOLVEMENT BY LYMPHOMA: Platelets ≥ 75,000/mm^3. NOTE: Platelet transfusions are not permitted within 7 days of platelet assessment unless cytopenia is secondary to disease involvement
* WITH BONE MARROW INVOLVEMENT BY LYMPHOMA AND/OR DISEASE-RELATED CYTOPENIAS: Platelets ≥ 50,000/mm^3. NOTE: Platelet transfusions are not permitted within 7 days of platelet assessment unless cytopenia is secondary to disease involvement
* Hemoglobin ≥ 8 g/dL. NOTE: Red blood cell transfusions are not permitted within 7 days of hemoglobin assessment unless cytopenia is secondary to disease involvement
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN). If hepatic involvement by lymphoma, or Gilbert's disease: ≤ 3 x ULN
* Aspartate aminotransferase (AST) ≤ 2.5 x ULN. If hepatic involvement by lymphoma: AST ≤ 5 x ULN
* Alanine aminotransferase (ALT) ≤ 2.5 x ULN. If hepatic involvement by lymphoma: ALT ≤ 5 x ULN
* Creatinine clearance of ≥ 40 mL/min per 24 hour urine test or the Cockcroft-Gault formula
* IF NOT RECEIVING ANTICOAGULANTS: International normalized ratio (INR) OR prothrombin (PT) ≤ 1.5 x ULN
* IF ON ANTICOAGULANT THERAPY: PT must be within therapeutic range of intended use of anticoagulants
* IF NOT RECEIVING ANTICOAGULANTS: Activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN
* IF ON ANTICOAGULANT THERAPY: aPTT must be within therapeutic range of intended use of anticoagulants
* WOMEN OF CHILDBEARING POTENTIAL (WOCBP): Negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females of childbearing potential to abstain from heterosexual intercourse or use two adequate method of birth control, including at least 1 method with a failure rate of < 1% per year, for at least 28 days prior to day 1 of cycle 1, during the treatment period (including periods of treatment interruption), until 3 months after the final dose mosunetuzumab, 3 months after the last dose of polatuzumab vedotin, and 3 months after the last dose of tocilizumab (if applicable). Women must refrain from donating eggs during this same period. Agreement by males to abstain from heterosexual intercourse or use a condom with female partners of childbearing potential or pregnant female partners during the treatment period and until 5 months after the last dose of polatuzumab vedotin, and 2 months after the last dose of tocilizumab (if applicable). Men must refrain from donating sperm during this same period

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only) with no identified cause other than menopause
  * Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, established proper use of hormonal contraceptives that inhibit ovulation, hormone releasing intrauterine devices, and copper intrauterine devices. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post-ovulation methods) and withdrawal are not acceptable methods of contraception

Exclusion Criteria:

* Prior treatment with mosunetuzumab or other CD20-directed bispecific antibodies. Prior exposure to 2 or less doses without evidence of resistance is allowed
* Prior treatment with polatuzumab vedotin or with an antibody-drug conjugate containing monomethyl auristatin E (MMAE). Prior exposure to 2 or less doses without evidence of resistance is allowed
* Allogeneic stem cell transplant within 2 years prior to day 1 of protocol therapy, requires immunosuppression, or has evidence of active-versus-host-disease

  * Patients who had an allogeneic transplant > 2 years prior to day 1 of protocol therapy must additionally have been stable off immunosuppressive agents for ≥ 2 months
* Autologous stem cell transplant within 100 days prior to day 1 of protocol therapy
* Chimeric antigen receptor (CAR)-T therapy within 30 days prior to day 1 of protocol therapy
* Prior use of any anti-lymphoma treatment with monoclonal antibody, radioimmunoconjugate or antineoplastic drug conjugate (ADC) within 4 weeks prior to day 1 of protocol therapy
* Treatment with any chemotherapeutic agent, or treatment with any other anti-cancer agent (investigational or otherwise) within 4 weeks or 5 half-lives of the drug, whichever is shorter, prior to day 1 of protocol therapy
* Treatment with radiotherapy within 2 weeks prior to day 1 of protocol therapy

  * If patients have received radiotherapy within 4 weeks prior to prior to day 1 of protocol therapy, patients must have at least one measurable lesion outside of the radiation field. Patients who have only one measurable lesion that was previously irradiated but subsequently progressed are eligible
* Live vaccine within 30 days prior to day 1 of protocol therapy
* Systemic immunosuppressive therapy (including, but not limited to, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [TNF] agents) with the exception of corticosteroid treatment for lymphoma symptom control must be tapered down to ≤ 10 mg/day prednisone or equivalent 14 days prior to day 1 of protocol therapy. Exceptions are:

  * Inhaled or topical steroids
  * Use of mineralocorticoids for management of orthostatic hypotension
  * Use of physiologic doses of corticosteroids for management of adrenal insufficiency
  * Use of 4 or less pulsed doses of steroids (i.e. dexamethasone) for urgent stabilization of lymphoma or symptom management
* Grade ≥ 2 peripheral neuropathy
* History of severe allergic or anaphylactic reaction to humanized, chimeric or murine monoclonal antibodies (or recombinant antibody-related fusion proteins)
* History of solid organ transplantation
* History of progressive multifocal leukoencephalopathy (PML)
* Known or suspected history of hemophagocytic lymphohistiocytosis (HLH)
* Significant active pulmonary disease (e.g., bronchospasm and/or obstructive pulmonary disease)
* Pneumonitis or interstitial lung disease requiring ongoing corticosteroid or immunosuppression and/or requirement for supplemental oxygen

  * Patients with any other history of pneumonitis or interstitial lung disease may be eligible after discussion with the study PI
* Positive severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) antigen or polymerase chain reaction (PCR) test within 7 days prior to day 1 of protocol therapy
* Clinically significant uncontrolled illness
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment or any major episode of infection requiring treatment with IV antibiotics or hospitalization (relating to the completion of the course of antibiotics) within 2 weeks prior to the first study treatment administration
* Known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection. Patients with past HBV infection (defined as negative hepatitis B surface antigen [HBsAg] and positive hepatitis B core antibody [HBcAb]) are eligible if HBV deoxyribonucleic acid (DNA) is undetectable. Patients who are positive for HCV antibody are eligible if PCR is negative for HCV ribonucleic acid (RNA). Testing to be done only in patients suspected of having infections or exposures
* Known active human immunodeficiency virus (HIV) infection. Subjects who have an undetectable or unquantifiable HIV viral load with CD4 > 200 and are on highly active antiretroviral therapy (HAART) medication are allowed. Testing to be done only in patients suspected of having infections or exposures
* Known or suspected chronic active Epstein-Barr virus (EBV) infection
* Known active central nervous system (CNS) involvement by lymphoma, including leptomeningeal involvement

  * Previously treated CNS involvement including disease with leptomeningeal involvement, is acceptable. Patients should be neurologically stable prior to study entry, and receiving a stable or decreasing corticosteroid dose
* History of CNS disease which was symptomatic or required treatment in the past 1 year, such as stroke, epilepsy, CNS vasculitis or neurodegenerative disease
* Symptomatic cardiac disease such as New York Heart Association class III or IV (including symptomatic ventricular dysfunction, symptomatic coronary artery disease, and symptomatic arrhythmias), cerebrovascular event/stroke or myocardial infarction within the past 6 months
* Clinically significant history of liver disease, including viral or other hepatitis, or cirrhosis
* Active autoimmune disease requiring systemic treatment
* History of autoimmune disease, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener granulomatosis, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis

  * Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone may be eligible
  * Patients with controlled type 1 diabetes mellitus who are on an insulin regimen are eligible for the study
  * Patients with a history of rheumatoid arthritis, Sjögren syndrome, systemic lupus erythematosus may be eligible after discussion with the study PI
  * Patients with a history of disease-related immune thrombocytopenic purpura, autoimmune hemolytic anemia, or other stable autoimmune diseases may be eligible after discussion with the study PI
* Recent major surgery (within 4 weeks) prior to start of protocol therapy, other than for diagnosis
* History of another primary malignancy that has not been in remission for at least 2 years, with the following exceptions:

  * Adequately treated non-melanoma skin cancer or lentigo maligna (melanoma in situ) without evidence of disease
  * Adequately treated in situ carcinomas (e.g. cervical, esophageal) without evidence of disease
  * Asymptomatic prostate cancer managed with a watch-and-wait strategy
  * If the malignancy is expected to not require any treatment for at least 2 years (this exception should be discussed with the study PI)
* Concomitant investigational therapeutic therapy or within 7 days prior to initiation of study treatment
* FEMALES ONLY: Pregnant or breastfeeding
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2028-03-14 (Estimated); Study Completion 2028-03-14 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 3 or higher adverse events (AEs) | Up to completion of first 2 cycles of treatment - each cycle is 28 days
  Unacceptable toxicity will be defined as events occurring during the first 2 cycles of treatment that is at least possibly related to study treatment. Observed toxicities will be summarized by type, severity, and attribution.
Complete response (CR) rate | Up to 36 months after last dose of protocol therapy
  CR rate will be defined as the proportion of response-evaluable participants that achieve a best response of CR after the start of protocol therapy and prior to disease progression and/or start of other anti-lymphoma therapy. CR rate will be estimated along with the 95% exact binomial confidence interval.

SECONDARY OUTCOMES:
Incidence of AEs | Up to 30 days from last dose of protocol therapy
  AEs will be graded by National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Cytokine release syndrome (CRS) will be graded according to the American Society for Transplantation and Cellular Therapy (ASTCT) CRS Consensus Grading Criteria. Immune Effector Cell Associated Neurotoxicity Syndrome (ICANS) will be graded according to the ASTCT ICANS Consensus Grading Criteria. Observed toxicities will be summarized by type, severity, and attribution.
Overall response rate (ORR) | Up to 36 months after last dose of protocol therapy
  ORR will be defined as the proportion of response-evaluable participants that achieve a best response of CR or partial response (PR) after the start of protocol therapy and prior to disease progression and/or start of other anti-lymphoma therapy. ORR will be estimated along with the 95% exact binomial confidence interval.
Time to first CR | At start of protocol therapy to CR up to 36 months after last dose of protocol therapy
  Time to first CR will be defined as the time from start of protocol therapy until the time the patients first achieve CR. Time for first CR will be summarized by descriptive statistics.
Time to best response | At start of protocol therapy to first best response up to 36 months after last dose of protocol therapy
  Time to best response will be defined as the time from start of protocol therapy until the time the patients achieve first best response (CR or PR). Time to best response will be summarized by descriptive statistics.
Duration of response (DOR) | At first PR or CR to progression or death up to 36 months after last dose of protocol therapy
  DOR will be defined as the time from first achievement of PR or CR to time of progression or death, whichever is earlier. DOR will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error. The 95% confidence interval will be constructed based on log-log transformation. Median DOR will be estimated when available.
Duration of response among CR (DORC) | At CR up to 36 months after last dose of protocol therapy
  DORC will be limited to patients who achieve a best response of CR. DORC will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error. The 95% confidence interval will be constructed based on log-log transformation.
Progression-free survival (PFS) | At start of protocol treatment to disease relapse/progression or death up to 36 months after last dose of protocol therapy
  PFS will be defined as the duration of time from start of protocol treatment to time of disease relapse or progression to death due to any cause, whichever occurs earlier. PFS will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error. The 95% confidence interval will be constructed based on log-log transformation. Median PFS will be estimated when available.
Overall survival (OS) | At start of protocol treatment to death up to 36 months after last dose of protocol therapy
  OS will be defined as the duration of time from start of protocol treatment to time of death due to any cause.OS will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error. The 95% confidence interval will be constructed based on log-log transformation. Median OS will be estimated when available.
Patient reported quality of life (QOL) | At baseline and up to 24 months of follow-up
  Patient reported QOL will be assessed using the European Quality of Life Five Dimension Five Level scale. Changes in QOL measures will be summarized by each timepoint and longitudinally.
Use of tocilizumab | Up to 36 months after last dose of protocol therapy
  Use of tocilizumab will be defined as the need to administer tocilizumab. Use of tocilizumab for CRS will be summarized by descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Mei, MD, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - City of Hope Orange County Lennar Foundation Cancer Center, Irvine, California